CLINICAL TRIAL: NCT01905358
Title: Title: The Study of Intra-articular Interventions of Platelet Rich Plasma or Hyaluronic Acid Compounds vs. Usual Care (Exercise/Diet/Supplements) in the Medical Management of Knee OA- Effects on Pain and Function; Effects on Articular Cartilage; Effects on Time to Partial or Total Knee Arthroplasty: The Knee Usual Care Evaluation (KUCE) Study
Brief Title: The Knee Usual Care Evaluation Study
Acronym: KUCE
Status: Terminated | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 29031
Record Dates: First submitted 2013-07-16; First posted 2013-07-23 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this prospective data collection is to track patients who are treated at HSS who are confirmed with knee osteoarthritis. The registry will collect prospective patient related and functional outcomes (including use of assistive devices), medication use and imaging data on patients with confirmed osteoarthritis, and the effect of different medical interventions that include PRP, Synvisc / Orthovisc /Euflexxa, bracing, suggested exercises, supplements, and diet. Information from the data collection will be used to compare outcomes of non-surgical alternatives with the end point being knee arthroplasty. The information results will enhance our knowledge of the long-term efficacy and effectiveness of non-surgical interventions intended to treat the progression of osteoarthritis.

Hypotheses:

* Different non-surgical interventions such as PRP, Synvisc®, Orthrovisc®, Euflexxa, bracing, physical therapy, and a prescribed combination of exercise, diet, and supplements will demonstrate statistically significant differences in patient pain and functional outcomes compared to usual interventions including use of NSAIDs, corticosteroid injections, and use of assistive devices such as canes.
* Non-operative interventions for knee osteoarthritis will be associated with different rates of breakdown of articular cartilage and different rates of progression of osteoarthritis as evidenced by MRI or joint space narrowing on standing knee films?
* Education about available non-operative treatment methods may change time the end point of total or partial knee replacement for patients with knee osteoarthritis of varying severity.
* Different non-operative interventions will be associated with different times to total or partial knee arthroplasty in patient with knee osteoarthritis of similar severity.
* An electronic data capture system (EDC) for osteoarthritis patients will improve patient care and patient outcomes.

DETAILED DESCRIPTION:
Specific Aims:

* To ascertain the long term success of non-surgical interventions intended to alleviate symptoms or slow progression of osteoarthritis of the knee.
* To ascertain if non-operative interventions for knee osteoarthritis improve patient pain, function, and quality of life.
* To ascertain if non-operative interventions for knee osteoarthritis affect the breakdown of articular cartilage and slow progression of osteoarthritis as evidenced by MRI or joint space narrowing on standing knee films?
* To ascertain the amount of time between the initial entry into care at HSS and the end point of total or partial knee replacement for patients with knee osteoarthritis of varying severity.
* To ascertain if non-operative interventions for knee osteoarthritis prolong time to knee replacement surgery.
* To implement at electronic data capture system (EDC) for osteoarthritis patients which will store validated patient reported outcomes, physical findings, and imaging results.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 30 years and less than 80 years
* Knee pain for at least 6 weeks
* Pain rate greater than or equal to 4/10 on a visual analog scale
* Morning stiffness less than 30 minutes
* Crepitus on active motion of the knee, bony tenderness, or bony enlargement of the knee
* Willing and able to consider all medical treatment options used to manage osteoarthritis of the knee
* No contraindications to knee radiographs or MRI
* Willing to participate in a registry
* Able to understand and sign a consent
* Able to answer registry questions independently

Exclusion Criteria:

* Diagnosis of a systemic rheumatic disease or crystalline arthritis (ie RA, SLE, systemic sclerosis, psoriatic arthritis or psoriasis, gout, pseudogout, lyme arthritis, reactive arthritis, viral arthritis
* pregnant or nursing
* unable to give informed consent
* contraindication to MRI such as indwelling paemaker or cochlear implant
* requirement of metal equipment (such as oxygen)
* known claustrophobia
* gadolinium allergy
* lack of fluency in English. Unfortunately, we do not have the financial resources to offer full translation services

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital for Special Surgery knee osteoarthritis patients
Sampling Method: Non-Probability Sample
Enrollment: 906 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03-21 (Actual); Study Completion 2014-03-21 (Actual)

PRIMARY OUTCOMES:
Short Form (12) Health Survey (SF-12) | 6 months, 12 months, 24 months, 36 months, 48 months and 60 months.
  Change is being assessed.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | 6 months, 12 months, 24 months, 36 months, 48 months and 60 months.
  Change is being assessed.

OTHER OUTCOMES:
Whole-Organ MRI Scoring (WORMS) | baseline, 1 year, 2 years, 5 years
  Changes in MRI will be measured by a chance in the Whole-Organ MRI Scoring (WORMS) score of femur and tibia, and Outerbridge score for cartilage. The Boston Osteoarthritis Knee Study defined cartilage loss using the WORMS score as "an increase in the score at any sub-region compared to baseline in any of the 14 subregions of the knee scored for cartilage in each knee." For patients who have only standing radiographs available a 0.7 mm loss of joint space will be considered a significant loss over 3 years. Bruyere et al predicted that "the cut off for minimum JSN maximizing sensitivity and specificity for predicting future surgery was a change of 0.7 mm or more in minimum joint space width over a period of three years." Note: change is being assessed.
X-ray with Kellgren-Lawrence Grading | baseline, 4 years
  Change is being assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Roos EM, Toksvig-Larsen S. Knee injury and Osteoarthritis Outcome Score (KOOS) - validation and comparison to the WOMAC in total knee replacement. Health Qual Life Outcomes. 2003 May 25;1:17. doi: 10.1186/1477-7525-1-17. PMID 12801417
- [Background] Peterfy CG, Guermazi A, Zaim S, Tirman PF, Miaux Y, White D, Kothari M, Lu Y, Fye K, Zhao S, Genant HK. Whole-Organ Magnetic Resonance Imaging Score (WORMS) of the knee in osteoarthritis. Osteoarthritis Cartilage. 2004 Mar;12(3):177-90. doi: 10.1016/j.joca.2003.11.003. PMID 14972335
- [Background] Cameron ML, Briggs KK, Steadman JR. Reproducibility and reliability of the outerbridge classification for grading chondral lesions of the knee arthroscopically. Am J Sports Med. 2003 Jan-Feb;31(1):83-6. doi: 10.1177/03635465030310012601. PMID 12531763
- [Background] Hunter DJ, Li J, LaValley M, Bauer DC, Nevitt M, DeGroot J, Poole R, Eyre D, Guermazi A, Gale D, Felson DT. Cartilage markers and their association with cartilage loss on magnetic resonance imaging in knee osteoarthritis: the Boston Osteoarthritis Knee Study. Arthritis Res Ther. 2007;9(5):R108. doi: 10.1186/ar2314. PMID 17958892
- [Background] Ornetti P, Brandt K, Hellio-Le Graverand MP, Hochberg M, Hunter DJ, Kloppenburg M, Lane N, Maillefert JF, Mazzuca SA, Spector T, Utard-Wlerick G, Vignon E, Dougados M. OARSI-OMERACT definition of relevant radiological progression in hip/knee osteoarthritis. Osteoarthritis Cartilage. 2009 Jul;17(7):856-63. doi: 10.1016/j.joca.2009.01.007. Epub 2009 Feb 9. PMID 19230857
- [Background] Lawrence RC, Helmick CG, Arnett FC, Deyo RA, Felson DT, Giannini EH, Heyse SP, Hirsch R, Hochberg MC, Hunder GG, Liang MH, Pillemer SR, Steen VD, Wolfe F. Estimates of the prevalence of arthritis and selected musculoskeletal disorders in the United States. Arthritis Rheum. 1998 May;41(5):778-99. doi: 10.1002/1529-0131(199805)41:53.0.CO;2-V. PMID 9588729
- [Background] Rhon D. Re: Zhang W, Moskowitz RW, Nuki G, et al. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage 2008;16:137-62. Osteoarthritis Cartilage. 2008 Dec;16(12):1585; author reply 1589. doi: 10.1016/j.joca.2008.04.019. Epub 2008 Jun 2. No abstract available. PMID 18515155
- [Background] Kon E, Mandelbaum B, Buda R, Filardo G, Delcogliano M, Timoncini A, Fornasari PM, Giannini S, Marcacci M. Platelet-rich plasma intra-articular injection versus hyaluronic acid viscosupplementation as treatments for cartilage pathology: from early degeneration to osteoarthritis. Arthroscopy. 2011 Nov;27(11):1490-501. doi: 10.1016/j.arthro.2011.05.011. Epub 2011 Aug 10. PMID 21831567
- [Background] Loza E, Benito-Ruiz P, Blanco F, de Miguel E, Roman JA; ARTROACAS study group, Spain. Feasibility and efficacy of a multidisciplinary health care programme for patients with knee osteoarthritis. Clin Exp Rheumatol. 2011 Nov-Dec;29(6):913-20. Epub 2011 Dec 22. PMID 22132760
- [Background] Keller SD, Bayliss MS, Ware JE Jr, Hsu MA, Damiano AM, Goss TF. Comparison of responses to SF-36 Health Survey questions with one-week and four-week recall periods. Health Serv Res. 1997 Aug;32(3):367-84. PMID 9240286
- [Background] Pincus T, Maclean R, Yazici Y, Harrington JT. Quantitative measurement of patient status in the regular care of patients with rheumatic diseases over 25 years as a continuous quality improvement activity, rather than traditional research. Clin Exp Rheumatol. 2007 Nov-Dec;25(6 Suppl 47):69-81. PMID 18021510
- [Background] Gourlay ML, Fine JP, Preisser JS, May RC, Li C, Lui LY, Ransohoff DF, Cauley JA, Ensrud KE; Study of Osteoporotic Fractures Research Group. Bone-density testing interval and transition to osteoporosis in older women. N Engl J Med. 2012 Jan 19;366(3):225-33. doi: 10.1056/NEJMoa1107142. PMID 22256806
- [Background] Roos EM, Roos HP, Lohmander LS. WOMAC Osteoarthritis Index--additional dimensions for use in subjects with post-traumatic osteoarthritis of the knee. Western Ontario and MacMaster Universities. Osteoarthritis Cartilage. 1999 Mar;7(2):216-21. doi: 10.1053/joca.1998.0153. PMID 10222220
- [Background] Poissant L, Pereira J, Tamblyn R, Kawasumi Y. The impact of electronic health records on time efficiency of physicians and nurses: a systematic review. J Am Med Inform Assoc. 2005 Sep-Oct;12(5):505-16. doi: 10.1197/jamia.M1700. Epub 2005 May 19. PMID 15905487
- [Background] Wilson AS, Kitas GD, Carruthers DM, Reay C, Skan J, Harris S, Treharne GJ, Young SP, Bacon PA. Computerized information-gathering in specialist rheumatology clinics: an initial evaluation of an electronic version of the Short Form 36. Rheumatology (Oxford). 2002 Mar;41(3):268-73. doi: 10.1093/rheumatology/41.3.268. PMID 11934962
- [Background] Spakova T, Rosocha J, Lacko M, Harvanova D, Gharaibeh A. Treatment of knee joint osteoarthritis with autologous platelet-rich plasma in comparison with hyaluronic acid. Am J Phys Med Rehabil. 2012 May;91(5):411-7. doi: 10.1097/PHM.0b013e3182aab72. PMID 22513879